CLINICAL TRIAL: NCT07045558
Title: HAIC in Combination With Atezolizumab Plus Bevacizumab as Conversion Therapy in Unresectable Hepatocellular Carcinoma: a Single-arm, Prospective Study
Brief Title: HAIC + Atezolizumab Plus Bevacizumab in Unresectable HCC
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2025-039-C
Record Dates: First submitted 2025-06-10; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Unresectable Hepatocellular Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental cohort: The experimental cohort is going to enroll unrescetable HCC patients, and they will receive HAIC in combination with atezolizumab plus bevacizumab as conversion therapy.

SUMMARY:
Patients with unresectable HCC will be enrolled in the cohort and will receive the combination therapy of HAIC and atezolizumab plus bevacizumab. The objective response rate is the primary endpoint, and the secondary endpoint includes disease control rate, conversion rate, pathologic complete response, major pathologic response, progression-free survival, recurrence-free survival, overall survival, quality of life, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 75 years old, with no gender restrictions.
2. Confirmed unresectable hepatocellular carcinoma (BCLC stage B/C) by histology, cytology, or clinical diagnosis.
3. At least one measurable lesion based on RECIST version 1.1.
4. Child-Pugh class A or B7.
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1.
6. No prior systemic therapy received, with an expected survival ≥12 weeks.
7. Adequate organ function meeting the following criteria:

   A. Hematological parameters (without blood transfusion within 14 days): Hemoglobin (Hb) ≥80 g/L, White blood cell count (WBC) ≥3 × 10⁹/L, Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L, Platelet count (PLT) ≥50 × 10⁹/L; B. Biochemical parameters: Total bilirubin (TBIL) <1.5 × upper limit of normal (ULN), Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <5 × ULN, Serum creatinine (Cr) ≤1.5 × ULN.
8. Contraception requirements: Women of childbearing age must have a negative serum or urine pregnancy test (HCG) within 7 days before enrollment and agree to use effective contraceptive methods during the trial period and for 8 weeks after the last dose. Men must either have undergone surgical sterilization or agree to use appropriate contraceptive methods during the trial period and for 8 weeks after the last dose.
9. Willingness to voluntarily participate in the study, with good compliance and commitment to follow-up.

Exclusion Criteria:

1. Known intrahepatic cholangiocarcinoma, mixed hepatocellular carcinoma, sarcomatoid HCC, or fibrolamellar carcinoma.
2. Concurrent autoimmune diseases, organ/hematopoietic stem cell transplantation history, or other malignancies.
3. Impaired consciousness, inability to cooperate with treatment, or active psychiatric disorders.
4. Transarterial chemoembolization (TACE), hepatic arterial infusion chemotherapy (HAIC), bevacizumab, molecular targeted therapy, atezolizumab, or other PD-1/PD-L1 inhibitors received before enrollment.
5. Major surgery, chemotherapy, radiotherapy, or systemic therapy for lesions received within 1 month before enrollment.
6. Use of immunosuppressants or systemic corticosteroids for immunosuppressive purposes (>10 mg/day prednisone or other equivalent drugs) within 14 days before enrollment.
7. Severe esophageal varices or high risk of bleeding assessed by endoscopy.
8. Evidence of decompensated liver function, including ascites, gastrointestinal bleeding, or hepatic encephalopathy.
9. Severe organ dysfunction in major organs such as the liver, kidneys, heart, lungs, or brain.
10. Other contraindications for interventional therapy, molecular targeted therapy, or immunotherapy.
11. Inability to undergo scheduled follow-up or concurrent participation in other clinical trials that may interfere with this study.
12. Other severe comorbidities deemed by the investigator to jeopardize patient safety or compromise study completion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who is diagnosed as unresectable hepatocellular carcinoma (BCLC stage B/C) histologically , cytologically, or clinically.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 2 years
  Complete response (CR) and partial response (PR), refer to cases evaluated by the mRECIST criteria for objective tumor response, including both CR and PR.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital affiliated to Shanghai Jiao Tong University, School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes